CLINICAL TRIAL: NCT05199805
Title: Mindfulness-Based Pain Management (MBPM) for Patients With Chronic Musculoskeletal Pain: a Randomized Controlled Trial.
Brief Title: Mindfulness-Based Pain Management (MBPM) for Patients With Chronic Musculoskeletal Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universität Duisburg-Essen (Other)
Responsible Party: Principal Investigator, Holger Cramer, PD Dr. rer. medic. Holger Cramer, Universität Duisburg-Essen
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 21-10081-BO
Record Dates: First submitted 2022-01-05; First posted 2022-01-20 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-12

CONDITIONS: Chronic Pain
Keywords: mindfulness; self-compassion; radnomized controlled trial
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Intervention Model Description: 40 patients with chronic (specific and non-specific) musculoskeletal pain will be randomized into two study conditions. The intervention group will receive MBPM sessions of 150 minutes each once a week for 8 weeks, while the control group will receive standard therapy (waiting list).
  The control group does not receive any active intervention in addition to treatment as usual during the intervention period. After completion of data collection, the control group will be offered an identical program, 6 months after randomization.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Data collectors will be blinded. Blinding of study participants is not possible due to the study design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-based pain management (Experimental): The program consists of sessions of 150 minutes once a week over the course of 8 weeks. Treatment as usual is allowed.
  Interventions: Behavioral: Mindfulness-based pain management
- Waiting-List (No Intervention): The control group will receive no active intervention in addition to treatment as usual during the study period.

INTERVENTIONS:
Behavioral: Mindfulness-based pain management — The structured program will include mindfulness exercises, meditation, a gentle body exercise series, and body awareness exercises, as well as information about pain, mindfulness-based pain management, and pain regulation methods suitable for everyday life. During the 8 weeks, treatment as usual is allowed.
  Other Names: Breathworks
  Arms: Mindfulness-based pain management

SUMMARY:
Mindfulness-Based Pain Management (MBPM) is an eight-week behavioral medicine program. Based on the well-known Mindfulness-Based Stress Reduction (MBSR) program, it was specifically developed as an intervention for chronic pain. During the program, mindfulness exercises, gentle body exercises and body awareness and breathing exercises, as well as pain regulation methods are taught.

Initial studies suggest efficacy of the program with regard to chronic pain, however, the effect of the standardized program in patients with chronic musculoskeletal pain has not yet been investigated in a clinical study. Therefore, the aim of this study is to investigate the MBPM program on pain acceptance in patients with chronic musculoskeletal pain. To this end, 40 patients with chronic (specific and non-specific) musculoskeletal pain will be randomly assigned to two study conditions. The intervention group will receive MBPM sessions of 150 minutes once a week over the course of 8 weeks, while the control group will receive standard therapy (waiting list). We hypothesize that patients will indicate a significantly higher pain acceptance after completing the program compared to patients not participating in the program.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the efficacy of a structured 8-week Mindfulness-Based Pain Management (MBPM) program, based on the Breathworks method by Vidyamala Burch, in addition to standard therapy compared to standard therapy alone in terms of pain acceptance in patients with chronic musculoskeletal pain.

The study is a monocentric, single-blinded (data collector), randomized study with 2 study arms. Study center is the Clinic for Natural and Integrative Medicine, Evang. Kliniken Essen-Mitte.

Patients will be recruited via study calls on the clinic website as well as via press advertisements (see appendix). In addition, former patients who have been treated at the Clinic for Natural and Integrative Medicine for chronic musculoskeletal pain will be contacted. If a patient reports interest in the study, he/she will first be screened by telephone for the presence of the inclusion and exclusion criteria. In case of potential eligibility, patients are invited to the Study Center. All patients will be informed by a study physician and assessed for suitability to participate in the study.

The inclusion and exclusion criteria are assessed on site by the study physician by means of a detailed general medical history and an orienting clinical-neurological examination.

Eligible patients will be assigned to one of the two study arms after completion of measurements at week 0 via non-stratified block randomization with randomly varying block length. Establishing the randomization sequence and ensuring blinded assignment will be done via central randomization through RedCap software by an external researcher who will have no patient contact throughout the study. Neither the patients nor the study physician nor the study coordinators will have any insight into the randomization sequence.

The study has 3 defined measurement time points: A baseline measurement (week 0) before randomization, at which time all standardized questionnaires as well as patient-specific data on sociodemographics (age, height, gender, weight, socioeconomic status), lifestyle, duration of disease, previous and currently applied therapies will be asked, and further measurement time points at the end of the course 8 weeks after randomization (week 8) and 6 months after randomization (week 26).

The sample size calculation was based on a non-randomized study by Cusens et al (2010), which found a large effect size of d=1.04 for pain acceptance for MBPM in addition to standard therapy compared to standard therapy alone. Based on a power (1-) of 80%, a significance level of 5%, and an anticipated dropout rate of up to 20%, a 2-sided t-test requires a total sample size of 40 patients (20 patients per group) to detect such an effect.

All analyses are based on the intention-to-treat population, i.e., all patients enrolled in the study are evaluated in the group originally assigned to them regardless of the treatment actually received. Missing values will be replaced using standard imputation procedures.

The primary outcome parameter will be analyzed confirmatively using univariate analysis of covariance (ANCOVA), in which the main outcome parameter will be modeled as a function of group membership (binary co-variate), respective baseline values (linear covariate), and expectancy (linear covariate). Within this model, the adjusted group difference (including 95% confidence interval) is estimated and tested for superiority of the intervention over the control group using a two-sided t-test at the α=0.05 level. Secondary end points will be evaluated exploratively using the same models as the primary end point. Change scores (change scores) and effect sizes (hedges' g) for between-group comparisons will be calculated to assess the clinical significance of the results.

The influence of potential process variables will be investigated using multiple mediator analyses.

ELIGIBILITY:
Inclusion Criteria:

- Chronic specific or nonspecific musculoskeletal pain for at least 3 months

Exclusion Criteria:

New diagnosis within the last 3 months of:

* Degenerative diseases (e.g., herniated disc, spinal stenosis)
* Neurological diseases (e.g., neuropathies, multiple sclerosis)
* Injuries of the spinal column (e.g. due to whiplash, vertebral body fractures, operations)

Or severe concurrent diagnosis of:

* Severe comorbid mental illness (e.g. addiction, severe depression)
* Severe comorbid physical illness (e.g. cancer diagnosis within the last 5 years, severe preexisting disease of the cardiovascular system, insufficiency of other organs (kidney, liver, etc.), acute febrile infection, other severe neurological diseases such as epilepsy)
* Pregnancy
* Current pension application (for work incapacity, occupational disability, reduction in earning capacity, severe disability)
* Simultaneous participation in other clinical trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-01-21 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-11-14 (Actual)

PRIMARY OUTCOMES:
pain acceptance | week 8
  Chronic Pain Acceptance Questionnaire, 20 items, range 0-6 with higher scores indicating a better outcome

SECONDARY OUTCOMES:
pain acceptance | week 26
  Chronic Pain Acceptance Questionnaire, 20 items, range 0-6 with higher scores indicating a better outcome
pain-associated self-efficacy | week 8 and 26
  Arthritis Self-Efficacy Scale, 9 items, range 1-10 with higher scores indicating a better outcome
pain intensity | week 8 and 26
  Numerical rating scale, range 0-10 with higher scores indicating a worse outcome
functional impairment | week 8 and 26
  pain disability index, 7 items, range 0-10 with higher scores indicating a worse outcome
health-related quality of life | week 8 and 26
  short form 12 with higher scores indicating a better outcome
psychiatric symptoms | week 8 and 26
  Hospital Anxiety and Depression Scale,14 items, range 0-3 with higher scores indicating worse outcomes

OTHER OUTCOMES:
mindfulness | week 8 and 26
  Conscious Presence and Self Control Scale, 10 items, range 0-3 with higher scores indicating a better outcome
self-compassion | week 8 and 26
  Self-Compassion Scale, 12 items, range 1-5 with higher scores indicating a better outcome
adverse events | week 8 and 26
  documentation by trainer
treatment expectancy | week 0
  Treatment Credibility Scale, 2 items, range 0-10 with higher scores indicating a better outcome
rationale credibility | week 8
  Treatment Credibility Scale, 3 items, range 0-10 with higher scores indicating a better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Holger Cramer, PhD, Principal Investigator — Universität Duisburg-Essen; Heidemarie Haller, PhD, Principal Investigator — Universität Duisburg-Essen
Locations (1):
- Universität Duisburg-Essen, Essen, Nordrhein-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cusens B, Duggan GB, Thorne K, Burch V. Evaluation of the breathworks mindfulness-based pain management programme: effects on well-being and multiple measures of mindfulness. Clin Psychol Psychother. 2010 Jan-Feb;17(1):63-78. doi: 10.1002/cpp.653. PMID 19911432